CLINICAL TRIAL: NCT00461201
Title: Effectiveness of an Intervention in Primary Care: Randomized Controlled Trial Comparing Care for Patients Requesting Same Day Consultations by Nurse Practitioner vs General Practitioners
Brief Title: Nurse vs General Practitioner Care for Patients Requesting Same Day Consultations in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catalan Institute of Health (Other Government)
Collaborators: Carlos III Health Institute (Other Government); Ministry of Health (Ambiguous); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PI060715
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2007-04-17 (Estimated); Status verified 2007-04

CONDITIONS: Acute Disease; Nursing Care; Ambulatory Care; Family Practice
Keywords: Health Services Research; Nurse Practitioners; Outcome and Process Assessment (Health Care); Patient Acceptance of Health Care; Patient Satisfaction; Primary Health Care; Professional Autonomy
MeSH Terms: conditions — Acute Disease; Patient Acceptance of Health Care; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Nurse practitioner care of patients

SUMMARY:
The purpose of this study is to compare the effectiveness of nursing care in relation to usual medical care in adult patients who demand to be visited the same day in Primary Care Teams in Catalonia, as it is suggested in other countries.

DETAILED DESCRIPTION:
The primary care demand is rapidly growing and the family physicians feel overflowed by the demand and their capacity to solve things is limited by lack of time. Many organizational interventions have been planned to solve this problem. One of these is to imply the nurse professional to solve and control health problems that traditionally were the doctor's job. So, to demonstrate the nursing care is as effective as the medical care, we will compare, among both collectives, the 'quality' of care received by patients who ask an appointment for the same day.

ELIGIBILITY:
Inclusion Criteria:

* patients requesting same day consultations in primary care
* assigned to the practice

Exclusion Criteria:

* do not want to participate
* difficulties to follow-up
* serious illness that makes the intervention impossible
* home visits

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1640
Dates: Start 2009-01

PRIMARY OUTCOMES:
Description of the capacity of resolution of the nurse:
To determine if there are differences in the proportion of patients that make a second appointment for the same reason in the next 2 weeks, comparing the two groups.
To determine if there are differences in the resolution of symptoms in 2 weeks after the visit comparing the two groups.
To determine if there are differences in the proportion of admission to hospital or to emergency room the next 2 weeks comparing the two groups.
To determine if there are differences in the satisfaction and resolution of the worries about the users state of health in 2 weeks after the visit comparing the two groups.
To determine if there are differences comparing the two groups in the perceived status of health, perception of the information, received attention, resource utilization and future intention to consult again with the same professional.

SECONDARY OUTCOMES:
Description of the clinical demands of the users and their demographic characteristics.
To identify if there is a type of user in which the effectiveness of the intervention is higher.
To determine the proportion of users visited by the nurse not having to be visited by the doctor afterwards for that reason.

CONTACTS AND LOCATIONS:
Overall Officials: Begoña Iglesias, Physician, Principal Investigator — Catalan Institute of Health; Maria Teresa Grifell, Nurse, Study Chair — Catalan Institute of Health; Josep Maria Vidal, Physician, Study Chair — Catalan Institute of Health; Sandra Pons, Physician, Study Chair — Catalan Institute of Health; Josep Casajuana, Physician, Study Chair — Catalan Institute of Health; Rosa Aragonès, Physician, Study Chair — Catalan Institute of Health; Mireia Fàbregas, Physician, Study Chair — Catalan Institute of Health; Neus Esgueva, Nurse, Study Chair — Catalan Institute of Health; Anna Calvet, Physician, Study Chair — Catalan Institute of Health; Maria Teresa Duran, Nurse, Study Chair — Catalan Institute of Health; Cristina Gallardo, Pysician, Study Chair — Catalan Institute of Health; Maria Assumpció Jiménez, Nurse, Study Chair — Catalan Institute of Health; Francisca Ramos, Physician, Study Chair — Catalan Institute of Health; Pere Joan Cortés, Physician, Study Chair — Catalan Institute of Health; Maria José Garcia, Physician, Study Chair — Catalan Institute of Health; Amparo Romaguera, Physician, Study Chair — Catalan Institute of Health; Soledad Romea, Physician, Study Chair — Catalan Institute of Health; Hèlia Cebrián, Nurse, Study Chair — Catalan Institute of Health; Jeannine Hernández, Physician, Study Chair — Catalan Institute of Health; Ramon Morera, Physician, Study Chair — Catalan Institute of Health; Manel Ferran, Physician, Study Chair — Catalan Institute of Health; Isabel Rosich, Farmacy, Study Chair — Catalan Institute of Health; Maria Carmen Sanchez, Nurse, Study Chair — Catalan Institute of Health

REFERENCES:
- [Background] Effectiveness of health checks conducted by nurses in primary care: final results of the OXCHECK study. Imperial Cancer Research Fund OXCHECK Study Group. BMJ. 1995 Apr 29;310(6987):1099-104. PMID 7742676
- [Background] Mundinger MO, Kane RL, Lenz ER, Totten AM, Tsai WY, Cleary PD, Friedewald WT, Siu AL, Shelanski ML. Primary care outcomes in patients treated by nurse practitioners or physicians: a randomized trial. JAMA. 2000 Jan 5;283(1):59-68. doi: 10.1001/jama.283.1.59. PMID 10632281
- [Background] Kinnersley P, Anderson E, Parry K, Clement J, Archard L, Turton P, Stainthorpe A, Fraser A, Butler CC, Rogers C. Randomised controlled trial of nurse practitioner versus general practitioner care for patients requesting "same day" consultations in primary care. BMJ. 2000 Apr 15;320(7241):1043-8. doi: 10.1136/bmj.320.7241.1043. PMID 10764366
- [Background] Venning P, Durie A, Roland M, Roberts C, Leese B. Randomised controlled trial comparing cost effectiveness of general practitioners and nurse practitioners in primary care. BMJ. 2000 Apr 15;320(7241):1048-53. doi: 10.1136/bmj.320.7241.1048. PMID 10764367
- [Background] Shum C, Humphreys A, Wheeler D, Cochrane MA, Skoda S, Clement S. Nurse management of patients with minor illnesses in general practice: multicentre, randomised controlled trial. BMJ. 2000 Apr 15;320(7241):1038-43. doi: 10.1136/bmj.320.7241.1038. PMID 10764365
- [Background] Horrocks S, Anderson E, Salisbury C. Systematic review of whether nurse practitioners working in primary care can provide equivalent care to doctors. BMJ. 2002 Apr 6;324(7341):819-23. doi: 10.1136/bmj.324.7341.819. PMID 11934775
- [Background] Zwarenstein M, Bryant W. Interventions to promote collaboration between nurses and doctors. Cochrane Database Syst Rev. 2000;(2):CD000072. doi: 10.1002/14651858.CD000072. PMID 10796485